CLINICAL TRIAL: NCT06738797
Title: Evaluation de l'Association Entre Les résultats d'un Test in Vitro en Cours de développement (SPHERTEST) et la réponse Aux Traitements Par Inhibiteur du Point de contrôle Chez Des Patients Atteints de Carcinome urothélial de Stade avancé ou métastatique.
Brief Title: Association Between the SPHERTEST in Vitro Test and Response to Checkpoint Inhibitor Treatments in Patients With Advanced or Metastatic Urothelial Carcinoma
Acronym: PROMES-URO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-2/NH01
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Urogenital Neoplasms
MeSH Terms: conditions — Urogenital Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood sampling (5 EDTA tubes of 4 ml or 20 ml in total) before and after initiation of immunotherapy.
  Stool sampling at the patient's home using a dedicated kit before starting immunotherapy and then before cycle 4 ( of treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with urothelial carcinoma
  Interventions: Diagnostic Test: SPHERTEST test

INTERVENTIONS:
Diagnostic Test: SPHERTEST test — The SPHERETEST is an in vitro model of heterotypic spheroids composed of commercial urothelial carcinoma tumor cells and leukocyte mononuclear cells from healthy donors.

SUMMARY:
First-line systemic treatments for bladder cancer are based on a combination of cytotoxic and immunotherapy, sequentially or concomitantly. Immune checkpoint inhibition (ICPI) is a powerful treatment for patients with metastatic urothelial carcinoma (UC). Since 2017, pembrolizumab (anti-PD1) can be offered as a second-line treatment after failure of platinum agents. In patients responding to platinum salts in first-line treatment, it is possible to maintain efficacy with maintenance treatment with another ICPI, avelumab (anti-PDL1). The phase III JAVELIN BLADDER 100 study compared avelumab to supportive care alone after successful platinum-based chemotherapy. At 30 months, 19.3% of patients were still in response compared to only 6.3% in the supportive care arm. However, biomarker analysis on tumor tissue did not show a robust signature on an individual scale. Recently, two phase 3 trials in first-line were presented at the ESMO 2023 congress. The first, in patients who could receive cisplatin-based chemotherapy, found a benefit on overall survival of adding Nivolumab in combination and then maintaining it for two years. The second proposed combined Enfortumab Vedotin and Pembrolizumab versus standard chemotherapy, with an overall survival for the study arm of more than 31 months. These trials confirm the essential role of immunotherapy in urothelial carcinomas. This progress is tempered by toxicity, cost and the lack of data on patient selection and treatment sequence. Although "prognostic" biomarkers have been identified, they cannot guide the choice of therapy, but only predict the expected outcomes, regardless of the treatment; biomarkers capable of predicting clinical benefit ("predictive") are urgently needed. It is therefore essential to identify a predictive signature at the individual level. The study authors have validated an in vitro model of heterotypic spheroids (SPHERTEST) composed of commercial urothelial carcinoma tumor cells and PBMCs from healthy donors. The aim of the study is to validate this model with PBMCs from UC patients to evaluate the effects of immunotherapy on the immune response and on tumor cell survival in vitro.

The study hypothesis is that the outcome of the pre-therapeutic test based on a heterotypic spheroid model with PBMC from patients with advanced or metastatic urothelial carcinoma (SPHERTEST) is related to the response to checkpoint inhibitor (CI) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven urothelial carcinoma, in a locally advanced or metastatic situation with indication for immunotherapy.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in a category 1 or drug monotherapy interventional study, or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* History of treatment with anti-PD1 or anti-PDL1 or anti-CTLA4 within the year.
* Pregnant, parturient or breastfeeding patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with advanced or metastatic urothelial carcinoma with an indication for treatment with an immune checkpoint inhibitor treated in the onco-urology departments of the Nîmes University Hospitals, the Antoine Lacassagne Center, the IUCT Toulouse and the Montpellier Regional Cancer Institute.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
SPHERTEST measurement of potential therapeutic efficacy | Day 0
  Yes/No. Differential in spheroid size before and after treatment according to the formula: R=M1-M0. R = test results, M0 = average spheroid size without immunotherapy treatment, M1 = average spheroid size with immunotherapy treatment. When R is ≤ 0, SPHERTEST = "yes" or "potential therapeutic efficacy". When R is > 0, SPHERTEST = "no" or "absence of potential therapeutic efficacy"
Progression-free survival | Month 12
  Yes/No according to RECIST criteria

SECONDARY OUTCOMES:
Histology of cells | Inclusion
  Pure transitional cells vs predominantly transitional cells
Presence of an aggressive minority component | Inclusion
  Yes/no
Type of other component | Inclusion
  Micropapillary, microcystic, trophoblastic differentiation, epidermoid differentiation, nested, plasmacytoid, sarcomatoid, rhabdoid, lymphoepitheliomatoid, large cell, undifferentiated or neuroendocrine
Tumor grade | Inclusion
  WHO grading
PD1/PDL1 status | Inclusion
  Yes/no
PDL1 score | Inclusion
  positive/negative
Type of metastatic involvement | Inclusion
  Locally advanced (= local recurrence, or pelvic lymph node involvement) or Metastatic sites: liver, bone, lung, brain, extrapelvic lymph node, other
Primary tumor site | Inclusion
  Bladder/Urethra/upper urinary tract/Urethra
Hemoglobin level | Inclusion
  g/dL
Hemoglobin level | Cycle 2 visit
  g/dL
Lactate dehydrogenase level | Inclusion
  UI/L
Lactate dehydrogenase level | Cycle 2 visit
  UI/L
C-reactive protein level | Inclusion
  mg/L
C-reactive protein level | Cycle 2 visit
  mg/L
Neutrophil count | Inclusion
  G/L
Neutrophil count | Cycle 2 visit (cycles are spaced 3 weeks (pembrolizumab) or 2 weeks (avelumab) apart)
  G/L
Lymphocyte count | Inclusion
  G/L
Lymphocyte count | Cycle 2 visit (cycles are spaced 3 weeks (pembrolizumab) or 2 weeks (avelumab) apart)
  G/L
Number of lines of systemic treatment received in the metastatic phase | Inclusion
  0, 1, 2, ≥3
Type of platinum salt received prior to immunotherapy | Inclusion
  Cisplatin or carboplatin
Treatment regimen prior to anti-PD1 therapy | Inclusion
  Neoadjuvant with progression within 12 months / Adjuvant with progression within 12 months / Initially locally advanced/metastatic
Current treatment: whether treatment is combined with another molecule | Inclusion
  Cisplatin / entoftumab-vedotin
Antibiotics in the previous month | Inclusion
  Duration (days)
Corticosteroid therapy > 10 mg prednisolone equivalent at immunotherapy initiation | Inclusion
  Yes/no
Taking an immunosuppressant other than corticosteroid therapy at immunotherapy initiation | Inclusion
  Yes/no
Any comedication at immunotherapy initiation | Inclusion
  Protein pump inhibitors / beta blockers / metformin / statin
Patient functioning level | Inclusion
  ECOG Performance Status Scale (1-5)
BCG vaccine | Inclusion
  Yes/no
Mitomycin therapy | Inclusion
  Yes/no
History of auto-immune disease | Inclusion
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Houede, Principal Investigator — CHU de Nimes
Locations (5):
- France (5):
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CHU de Nimes, Nîmes
  - Iuct Oncopole, Toulouse